CLINICAL TRIAL: NCT07396324
Title: NEOadjuvant Iparomlimab and Tuvonralimab (QL1706) Plus Chemotherapy in Patients With Hormone Receptor Positive And HER2-Negative Breast Cancer: a Prospective, Single Arm, Multicenter Clinical Trial
Brief Title: Neoadjuvant Iparomlimab and Tuvonralimab (QL1706) in Patients With Hormone Receptor Positive, HER2-negative Breast Cancer
Acronym: NEO-ITHRAN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY2025-422-A
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Hormone Receptor Positive/Human Epidermal Growth Factor Receptor 2 Negative Breast Cancer
MeSH Terms: interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant Iparomlimab and Tuvonralimab (QL1706) (Experimental): Iparomlimab and Tuvonralimab (QL1706) in combination with weekly paclitaxel and carboplatin as neoadjuvant therapy
  Interventions: Drug: Iparomlimab and Tuvonralimab (QL1706); Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab (QL1706) — 5.0mg/kg qw, start from C1D15
Drug: Paclitaxel — 80mg/m^2 qw
Drug: Carboplatin — AUC=1.5, D1, 8, 15, every 28 days

SUMMARY:
This is an prospective, open label, multicenter study to evaluate the efficacy and safety of neoadjuvant Iparomlimab and Tuvonralimab (QL1706) in patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Histologically confirmed hormone receptor positive and human epidermal growth factor receptor 2 (HER2) negative breast cancer
* Subjects with at least one evaluable lesion
* ECOG 0-1
* Adequate organ function

Exclusion Criteria:

* Metastatic disease (Stage IV)
* Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test;Female patients of childbearing age that are reluctant to take effective contraceptive measures throughout the trial period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with pCR | 1-2 weeks after surgery
  Number of patients with pathological complete response/Number of all eligible patients

SECONDARY OUTCOMES:
Proportion of patients with adverse events | From the date of starting neoadjuvant therapy to the end of the treatment (up to approximately 1 year)
  Number of patients with adverse events during neoadjuvant therapy assessed according to the NCI CTCAE v5.0/Number of all eligible patients

CONTACTS AND LOCATIONS:
Overall Officials: Wenjin Yin, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided